CLINICAL TRIAL: NCT04612205
Title: Effect of TECAR in Treating Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: eman elhosary (Other)
Responsible Party: Sponsor-Investigator, eman elhosary, assist .Prof.of women health department, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tecar & stress incontinence
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence, TECAR
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): females complain from SUI treated by TECAR and pelvic floor exercises
  Interventions: Device: TECAR followed by pelvic floor exercises
- group B (Active Comparator): females treated by pelvic floor exercises only
  Interventions: Other: pelvic floor exercises

INTERVENTIONS:
Device: TECAR followed by pelvic floor exercises — The signal generator was an INDIBA® 448 kHz RF device (vagina/rectum) (INDIBA SA, Barcelona, Spain).
  Arms: group A
Other: pelvic floor exercises — The patients will instructed to contract their pelvic floor muscles without contracting adjacent muscles, such as the abdomen, glutei and hip adductors muscles twenty repletion consisted of contraction and squeezing of the muscle ten seconds followed by relaxation for twenty second then rested for two minutes. The exercises program lasted for lasting 45 min. divided into 5 min. warming up, 35 min. actual treatment and 5 min. cooling down, three times a week for eight consecutive weeks. The patient will teach to contract their pelvic floor muscles before coughing or sneezing thus to prevent leakage. Home exercises through continuing practicing these contractions as frequent as possible according to her ability, at early morning before getting from bed from crock lying position, at afternoon from sitting and standing positions, at evening from sitting and standing positions and finally at night at bed time from crock lying position.
  Arms: group B

SUMMARY:
Stress urinary incontinence (SUI) is the defined as a leakage of urine with physical exertion, most commonly from coughing, laughing, or sneezing. It has a profound psychosocial impact not only to patients but also on their families and caregivers, resulting in loss of self stem, sexual dysfunction.Because of the higher incidence of stress urinary incontinence that reach 30% of women during childbearing period, 50% in elderly women, and its social embarrassing condition causing socio-psychological problems, disability and dependency with higher economic impact and based on TECAR therapy had better recovery of muscle strength and function in addition to there is no study has evaluated the impact of TECAR treatment on stress urinary incontinence, our study aim to assess the effectiveness of TECAR in treatment of such cases to decrease time of treatment and provide good results to patients.

ELIGIBILITY:
Inclusion Criteria:Participants aged between30 to 50 year and BMI not exceed 30 kg/cm2. All subjects complain from mild SUI due to hypermobility of bladder neck and weakness of pelvic floor exercise

-

Exclusion Criteria:

* Those with neurological diseases, diabetic neuropathy, congenital urologic disease, bladder cancer and neurogenic bladder, detrusor hyperactivity and bladder or urethra previous surgery

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
strength of pelvic floor | after 4 week
  strength of pelvic floor muscles measured by perineometer before treatment and after 4 weeks

SECONDARY OUTCOMES:
severity of SUI | after 4 weeks
  measured by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: eman elhosary, Principal Investigator — kafr elshekh university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elhosary EA, Ahmed Hamada H, Ali AlMubali F, Lopez Sanchez GF, Ahmed SM. Effect of monopolar capacitive resistive radiofrequency in treating stress urinary incontinence: A pilot randomized control trial. Front Psychol. 2023 Jan 5;13:1062363. doi: 10.3389/fpsyg.2022.1062363. eCollection 2022. PMID 36687887